CLINICAL TRIAL: NCT05094609
Title: Phase 1, Open Label Study to Evaluate the Safety and Immunogenicity of ChAd68 and AdHu5 Vector-based Trivalent COVID-19 Vaccines Delivered Via Inhaled Aerosol
Brief Title: Phase 1 Trial of ChAd68 and Ad5 Adenovirus COVID-19 Vaccines Delivered by Aerosol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M010
Record Dates: First submitted 2021-10-25; First posted 2021-10-26 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: COVID-19; SARS-CoV2 Infection
Keywords: COVID-19; SARS-CoV-2; Aerosol; Adenovirus; Chimpanzee; Immunogenicity; Inhalation; Vaccine; Vaccination
MeSH Terms: conditions — COVID-19; Adenoviridae Infections; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Dose escalation: Assuming no safety signal, the dose for each vaccine (Ad5-triCoV/Mac and ChAd-triCoV/Mac) will be escalated from a dose of 10e5 TCID50/dose (n=3/vaccine group), to a dose of 10e6 (n=3/vaccine group) and then further increased for each vaccine group to 1x10e7 (n=3 per group) and 3x10e7 (n=3 per group) assuming no safety signal. Based on poor immune responses to Ad5-triCoV/Mac the dose of Ad5-triCoV/Mac will not be further escalated. Since immunogenicity endpoints were not met at 3x10e7 for ChAd-triCoV/Mac and there was no safety signal, the dose will be further escalated to 6x10e7 and 1x10e8 (n=3 per dose level). Participants with a history of COVID infection will be enrolled to receive ChAd-triCoV/Mac, beginning with a dose of 3x10e7 (n=3) and, in the absence of any safety signal, escalated to 6x10e7 and, if required, 1x10e8 and, once the optimal dose has been determined, participants enrolled at this dose level to complete enrolment of the cohort (n=6).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Aerosol Ad5-triCoV/Mac dose level 10e5 (Experimental): Single dose by inhalation of 10e5 Ad5-tri-CoV/Mac
  Interventions: Biological: Ad5-triCoV/Mac
- Aerosol ChAd-tri-CoV/Mac dose level 10e5 (Experimental): Single dose by inhalation of 10e5 ChAd-triCoV/Mac
  Interventions: Biological: ChAd-triCoV/Mac
- Aerosol Ad5-triCoV/Mac dose level 10e6 (Experimental): Single dose by inhalation of 10e6 Ad5-triCoV/Mac
  Interventions: Biological: Ad5-triCoV/Mac
- Aerosol ChAd-triCoV/Mac dose level 10e6 (Experimental): Single dose by inhalation of 10e6 ChAd-triCoV/Mac
  Interventions: Biological: ChAd-triCoV/Mac
- Aerosol Ad5-triCoV/Mac dose level 10e7 (Experimental): Single dose by inhalation of 10e7 Ad5-triCoV/Mac
  Interventions: Biological: Ad5-triCoV/Mac
- Aerosol ChAd-triCoV/Mac dose level 10e7 (Experimental): Single dose by inhalation of 10e7 ChAd-triCoV/Mac
  Interventions: Biological: ChAd-triCoV/Mac
- Aerosol Ad5-triCoV/Mac dose level 3x10e7 (Experimental): Single dose by inhalation of 3x10e7 Ad5-triCoV/Mac
  Interventions: Biological: Ad5-triCoV/Mac
- Aerosol ChAd-triCoV/Mac dose level 6x10e7 (Experimental): Single dose by inhalation of 6x10e7 ChAd-triCoV/Mac
  Interventions: Biological: ChAd-triCoV/Mac
- Aerosol ChAd-triCoV/Mac dose level 1x10e8 (Experimental): Single dose by inhalation of 1x10e8 ChAd-triCoV/Mac
  Interventions: Biological: ChAd-triCoV/Mac
- ChAd-triCoV/Mac at a dose level of 3x10e7 (Experimental): Single dose by inhalation of 3x10e7 Ad5-triCoV/Mac
  Interventions: Biological: ChAd-triCoV/Mac

INTERVENTIONS:
Biological: Ad5-triCoV/Mac — Ad5-triCoV/Mac is a recombinant type 5 human adenovirus vector which has been engineered to express our trivalent SARS-CoV-2 transgene cassette under the control of an MCMV promoter, and is followed by an SV40 polyA signal. The adenovirus construct is E1 and E3 deleted.This trivalent transgene cassette consists of the S1 region of SARS-CoV-2 spike protein (aa 47-716), full-length SARS-CoV-2 nucleoprotein (N) fused to a highly conserved portion of the SARS-CoV-2 polymerase (RdRp or POL).
  Arms: Aerosol Ad5-triCoV/Mac dose level 10e5; Aerosol Ad5-triCoV/Mac dose level 10e6; Aerosol Ad5-triCoV/Mac dose level 10e7; Aerosol Ad5-triCoV/Mac dose level 3x10e7
Biological: ChAd-triCoV/Mac — ChAd-triCoV/Mac is an E1 and E3 deleted chimpanzee adenovirus serotype 68 where the trivalent SARS-CoV-2 transgene cassette is under the control of an HCMV promoter and is followed by an SV40 polyA signal. The trivalent transgene cassette consists of the S1 region of SARS-CoV-2 spike protein (aa 47-716), full-length SARS-CoV-2 nucleoprotein (N) fused to a highly conserved portion of the SARS-CoV-2 polymerase (RdRp or POL).
  Arms: Aerosol ChAd-tri-CoV/Mac dose level 10e5; Aerosol ChAd-triCoV/Mac dose level 10e6; Aerosol ChAd-triCoV/Mac dose level 10e7; Aerosol ChAd-triCoV/Mac dose level 1x10e8; Aerosol ChAd-triCoV/Mac dose level 6x10e7; ChAd-triCoV/Mac at a dose level of 3x10e7

SUMMARY:
This is a phase 1 study in healthy volunteers who have received at least three doses of an mRNA COVID-19 vaccine, to evaluate the safety and immune responses that develop in the blood and lungs following the administration by aerosol of either Ad5-triCoV/Mac or ChAd-triCoV/Mac, new experimental adenovirus-based vaccines expressing SARS-CoV-2 spike, nucleocapsid and RNA polymerase proteins.

DETAILED DESCRIPTION:
This is a phase 1, dose-escalating study to evaluate the safety and immunogenicity of a single dose of either Ad5-triCoV/Mac, a replication deficient human adenovirus vector, or ChAd-triCoV/Mac, a replication deficient chimpanzee adenovirus 68 vector, delivered to the respiratory tract by aerosol, in healthy volunteers who have received at least three doses of an mRNA COVID-19 vaccine. Both vectors have been engineered to express the spike, nucleocapsid and RNA polymerase proteins.

Up to 36 healthy volunteers will be enrolled in this dose escalation study. The first cohort (n=6) will receive Ad5-triCoV/Mac (n=3) or ChAd-triCoV/Mac (n=3) at the lowest dose of 10e5 TCID50, administered using the AeroNeb Solo Vibrating Mesh Nebulizer. Assuming no safety concerns, participants will then be administered Ad5-triCoV/Mac (n=3) or ChAd-triCoV/Mac (n=3) at a dose of 10e6. Assuming no safety signals we will move to vaccinate at the next dose level of 1x10e7 TCID50. Decisions about dose escalation will be made independently for each vaccine based on safety and immunogenicity profile. If the immunogenicity endpoints are not reached, in the absence of a safety signal, at the 10e7 dose level, we will move to the next dose level of 3x10e7 TCID50 and enrol three participants/vaccine group. Similarly, if all of the immunogenicity endpoints in the BAL are not met at 3x10e7, and in the absence of any safety signal, we will further escalate to 6x10e7, then 1x10e8 TCID50 and enrol three participants/vaccine group, if required. Once safety has been shown in participants without a history of COVID, we will proceed to enrol participants with a history of COVID infection to receive ChAd-triCoV/Mac, beginning with a dose of 3x10e7 (n=3) and, in the absence of any safety signal, escalating to 6x10e7 and, if required, 1x10e8 and, once the optimal dose has been determined based on immunogenicity outcomes, continue to enrol participants at this dose level to complete enrolment of the cohort (n=6).

Antibody and specific T cell responses will be measured in lung from bronchoalveolar lavage fluid collected at bronchoscopy at baseline and at 4 weeks following vaccination and in blood at several time points up to week 48 following vaccination.

Safety endpoints will include the nature of any adverse events, their severity and the probability of a relationship to study procedures and administration of vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy human subjects who are between 18 and 65 years of age.
2. Have completed a COVID vaccine series with at least three doses of a licensed mRNA vaccine at least 3 months prior.
3. HIV antibody negative.
4. Able to understand and comply with protocol requirements and instructions; able to attend scheduled study visits and complete required investigations.
5. For women, negative pregnancy test and for those women of child-bearing potential practising two acceptable forms of contraception for the duration of the study.
6. For men, using barrier contraception for the duration of the study.
7. No history of COVID infection OR history of documented COVID infection at least 6 months prior, dated from either a self-reported positive rapid antigen test or positive PCR test (self-reported or documented). For participants with a history of COVID infection, anti-nucleocapsid antibodies will be measured prior to enrolment to confirm infection.

Exclusion Criteria:

1. Subjects who have received any recombinant adenoviral-vectored COVID-19 vaccine, e.g. AstraZeneca COVISHIELD COVID-19 vaccine.
2. Pregnant or lactating women.
3. Subjects who have any acute or chronic illnesses, any relevant findings on physical examination or are receiving any immunosuppressive therapy in the opinion of the investigator likely to affect the immune system including current use of inhaled or nasal steroids.
4. Subjects with a history of any bleeding disorder or receiving any drug treatment that in the opinion of the investigator may increase the risk of bleeding.
5. Subjects with a history of respiratory diseases requiring regular treatment, e.g. asthma, COPD, interstitial lung diseases, bronchiectasis.
6. Current cigarette smokers, current e-cigarette smokers and ex-smokers who have quit less than a year ago, as reported by the subject.
7. Subjects with clinically significant abnormal baseline spirometry tests: FEV1<80% predicted, FVC<80% predicted, FEV1/FVC<70%; DLCO<70% predicted.
8. Any health-related condition for which study bronchoscopy is contraindicated.
9. Subjects whose baseline laboratory values are outside of the normal range, unless the abnormality is considered not clinically relevant by the investigator. A single repeat test is allowed during the screening period.
10. Subjects whose use of alcohol or drugs would, in the opinion of the investigator, interfere with adherence to the study protocol.
11. Subjects who are using, or have a history of using, inhaled cocaine, metamphetamine or other inhaled or smoked recreational drugs. Subjects who give a history of smoking marijuana more than a year ago may be enrolled as long as they agree not to smoke marijuana for the duration of the study.
12. Failure to provide written consent.
13. Known allergy to vaccine components.
14. Any abnormality on chest x-ray suggestive of clinically significant respiratory disease.
15. Previous receipt of any experimental adenovirus-vector vaccine by the aerosol route.
16. History of severe reaction to a previous COVID vaccination (including hives, difficulty breathing, angioedema, high fever, seizure).
17. History of venous or arterial thrombosis with thrombocytopenia following any vaccination.
18. History of cerebral venous thrombosis with thrombocytopenia.
19. History of heparin induced thrombocytopenia.
20. History of myocarditis or pericarditis.
21. History of Bell's Palsy.
22. History of hospitalization with an admitting diagnosis of primary COVID infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting adverse events and severity of adverse events following Ad5-triCoV/Mac vaccination | Over 48 weeks post vaccination
  Adverse events will be assessed according to the CTCAE Expanded Common Toxicity Criteria at 48-72 hours after vaccination, and at weeks 2, 4, 8, 12,16, 24, 32, 40 and 48
Number of participants reporting adverse events and severity of adverse events following ChAd-triCoV/Mac vaccination | Over 48 weeks post vaccination
  Adverse events will be assessed according to the CTCAE Expanded Common Toxicity Criteria at 48-72 hours after vaccination, and at weeks 2, 4, 8, 12,16, 24, 32, 40 and 48

SECONDARY OUTCOMES:
Immunogenicity of Ad5-triCoV/Mac administered by aerosol | Over 48 weeks post vaccination
  Change from baseline in: 1) spike-specific and anti-RBD antibodies including neutralizing antibodies both in the blood and airways; 2) spike/N/POL-specific CD4 and CD8 T cells in the airways (BAL fluid) four weeks post vaccination and 3) spike/N/POL-specific CD4 and CD8 T cells in the blood up to the last timepoint of examination.
Immunogenicity of ChAd-triCoV/Mac administered by aerosol | Over 48 weeks post vaccination
  Change from baseline in: 1) spike-specific and anti-RBD antibodies including neutralizing antibodies both in the blood and airways; 2) spike/N/POL-specific CD4 and CD8 T cells in the airways (BAL fluid) four weeks post vaccination and 3) spike/N/POL-specific CD4 and CD8 T cells in the blood up to the last timepoint of examination.
Immune response to Ad5-triCoV/Mac and ChAd-triCoV/Mac correlated with pre-existing adenovirus antibodies | Over 48 weeks
  Change from baseline in: 1) spike-specific and anti-RBD antibodies including neutralizing antibodies both in the blood and airways; 2) spike/N/POL-specific CD4 and CD8 T cells in the airways (BAL fluid) four weeks post vaccination and 3) spike/N/POL-specific CD4 and CD8 T cells in the blood up to the last timepoint of examination, correlated with baseline Ad5 antibodies
Correlation of antibodies measured in saliva with antibodies measured in BAL fluid and blood | Over 12 weeks
  Change from baseline in spike-specific and anti-RBD antibodies including neutralizing antibodies both in the blood and airways the airway (BAL fluid), correlated with antibodies measured in saliva

CONTACTS AND LOCATIONS:
Overall Officials: Fiona M Smaill, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
On request, individual patient data that underlie the results in a publication will be made to other researchers
Supporting Information: CSR
Time Frame: 3 months after publication
Access Criteria: Requests will be reviewed by the principal investigator and be judged on the scientific validity of the request and academic qualifications of those requesting access.

REFERENCES:
- [Background] Jeyanathan M, Afkhami S, D'Agostino MR, Satia I, Fritz DK, Miyasaki K, Ang JC, Zganiacz A, Howie KJ, Swinton M, Aguirre E, Zheng MB, Kazhdan N, Dvorkin-Gheva A, Mbuagbaw L, Medina MFC, Diab N, Brister DL, Gauvreau GM, Lichty BD, Miller MS, Smaill F, Xing Z. Induction of lung mucosal immunity by a next-generation inhaled aerosol COVID-19 vaccine: an open-label, multi-arm phase 1 clinical trial. Nat Commun. 2025 Jul 2;16(1):6000. doi: 10.1038/s41467-025-60726-0. PMID 40603330
- See also: Induction of lung mucosal immunity by a next-generation inhaled aerosol COVID-19 vaccine: an open-label, multi-arm phase 1 clinical trial — https://www.nature.com/articles/s41467-025-60726-0